CLINICAL TRIAL: NCT06236282
Title: Safety and Efficacy of Flexible Articulated Instrument (ArtiSential®) in Laparoscopic Surgery for Rectal Cancer
Brief Title: ArtiSential® for Rectal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2208-0071346
Record Dates: First submitted 2024-01-08; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ArtiSential® Use: Laparoscopic low anterior resection, with use of both straight devices and articulated devices
  Interventions: Device: ArtiSential®
- ArtiSential® Non-Use: Laparoscopic low anterior resection, with use of straight devices only

INTERVENTIONS:
Device: ArtiSential® — Articulated laparoscopic device made by Livsmed Co, South Korea.
  Groups: ArtiSential® Use

SUMMARY:
This study aimed to assess efficacy of ArtiSential® in reducing laparoscopic rectal cancer surgery duration. We retrospectively reviewed the data of patients who underwent laparoscopic low or ultralow anterior resection for primary mid-to-low rectal cancer, performed by a single surgeon in 2012-2022. Patients were divided into groups, use group vs. non-use group, based on the use or non-use of the ArtiSential®. The total mesorectal excision quality and resection margin status did not differ between the groups. ArtiSential® reduced operative time without impairing surgical quality or oncologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* mid-to-low rectal caner (witing 10cm of the anal verge)
* laparoscopic surgery

Exclusion Criteria:

* combined surgery
* recurrent rectal cancer surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent laparoscopic resection for mid-to low rectal cancer located within 10 cm of the anal verge, performed by a single experienced surgeon between 2012 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Operation time | 0 week
  To determine whether the use of articulated device can shorten total operative time

SECONDARY OUTCOMES:
Long-term Survival | 2 year
  2 year recurrence free survival and 2 year overall survival
Anastomotic leakage (postop outcome) | 4 weeks
  anastomotic leakage within one month
TME quality (Operative outcome) | 0 weeks
  Quality of total mesorectal excision to compare quality of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided